CLINICAL TRIAL: NCT00379041
Title: Protocol H8 for a Prospective Controlled Trial in Clinical Stage I-II Supradiaphragmatic Hodgkin's Disease. Evaluation of Treatment Efficacy and (Long Term) Toxicity in Three Different Prognostic Subgroups [H8 Trial]
Brief Title: Radiation Therapy With or Without Combination Chemotherapy in Treating Patients With Previously Untreated Stage I or Stage II Hodgkin's Lymphoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-20931; EORTC-20931-LYMG (Other: EORTC)
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; Doxorubicin; Mechlorethamine; Prednisone; Procarbazine; Vinblastine; Vincristine; Radiotherapy

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: doxorubicin hydrochloride
Drug: mechlorethamine hydrochloride
Drug: prednisone
Drug: procarbazine hydrochloride
Drug: vinblastine sulfate
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill cancer cells. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with combination chemotherapy may kill more cancer cells. It is not yet known whether radiation therapy is more effective with or without combination chemotherapy in treating patients with Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying radiation therapy to see how well it works with or without combination chemotherapy in treating patients with previously untreated stage I or stage II Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the efficacy of mantle field radiotherapy, in terms of overall survival, in patients with previously untreated stage I or II Hodgkin's lymphoma (HL) with a very favorable prognosis.
* Compare late treatment-related toxicity in patients with stage I or II HL with a favorable prognosis treated with standard subtotal nodal radiotherapy vs a combination of 3 courses of mechlorethamine, vincristine, procarbazine hydrochloride, prednisone/doxorubicin hydrochloride, bleomycin, and vinblastine (MOPP/ABV) followed by involved field radiotherapy.
* Compare overall survival and late treatment-related toxicity in patients with stage I or II HL with an unfavorable prognosis treated with 6 courses of MOPP/ABV followed by involved field radiotherapy vs 4 courses of MOPP/ABV followed by involved field radiotherapy vs subtotal nodal radiotherapy.
* Maintain the failure-free survival rate that was reached in previous studies, with a reduction of the acute side effects of the treatment, particularly severe late toxicity.

OUTLINE: This is a randomized, controlled, prospective, multicenter study. Patients are stratified according to prognosis (favorable vs unfavorable vs very favorable).

* Stratum 1 (very favorable prognosis): Patients undergo mantle field radiotherapy 5 days a week for at least 4 weeks.
* Stratum 2 (favorable prognosis): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients undergo subtotal nodal radiotherapy 5 days a week for at least 4 weeks.
  * Arm II: Patients receive mechlorethamine IV and vincristine IV on day 1; oral procarbazine hydrochloride on days 1-7; oral prednisone on days 1-14; and doxorubicin hydrochloride IV, bleomycin intramuscularly (IM) or IV, and vinblastine IV on day 8. Treatment repeats every 4 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Beginning 3-4 weeks after completion of chemotherapy, patients undergo involved field radiotherapy 5 days a week for at least 4 weeks.
* Stratum 3 (unfavorable prognosis): Patients are randomized to 1 of 3 treatment arms.

  * Arm I: Patients receive mechlorethamine IV and vincristine IV on day 1; oral procarbazine hydrochloride on days 1-7; oral prednisone on days 1-14; and doxorubicin hydrochloride IV, bleomycin IM or IV, and vinblastine IV on day 8. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Beginning 3-4 weeks after completion of chemotherapy, patients undergo involved field radiotherapy 5 days a week for at least 4 weeks.
  * Arm II: Patients receive chemotherapy as in arm I. Treatment repeats every 4 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo involved field radiotherapy as in arm I.
  * Arm III: Patients receive chemotherapy as in arm I. Treatment repeats every 4 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Beginning 3-4 weeks after completion of chemotherapy, patients undergo subtotal nodal radiotherapy 5 days a week for at least 4 weeks.

Quality of life is assessed after completion of study treatment and then annually for 10 years.

After completion of study treatment, patients are followed at 2, 4, 6, 9, and 12 months, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,158 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed supradiaphragmatic Hodgkin's lymphoma

  * Stage I or II disease
* Previously untreated disease

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Normal life expectancy
* No severe cardiac, pulmonary, neurologic, or metabolic disease that would interfere with normal life expectancy or study treatment
* No other prior or concurrent malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* No psychological, familial, socioeconomic, or geographic circumstance that would preclude proper staging or study compliance
* HIV negative
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior staging laparotomy
* No prior biologic therapy, chemotherapy, endocrine therapy, radiotherapy, or surgery for this malignancy

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1158 (Estimated)
Dates: Start 1993-09-01 (Actual); Primary Completion 1998-10-01 (Actual)

PRIMARY OUTCOMES:
Overall survival
Reduction of late treatment-related toxicity
Maintenance of failure-free survival rate

CONTACTS AND LOCATIONS:
Overall Officials: H. Eghbali, MD, Study Chair — Institut Bergonié; Christophe Ferme, Study Chair — Centre Medical de Bligny

REFERENCES:
- [Result] Heutte N, Flechtner HH, Mounier N, Mellink WA, Meerwaldt JH, Eghbali H, van't Veer MB, Noordijk EM, Kluin-Nelemans JC, Lampka E, Thomas J, Lugtenburg PJ, Viterbo L, Carde P, Hagenbeek A, van der Maazen RW, Smit WG, Brice P, van Marwijk Kooy M, Baars JW, Poortmans P, Tirelli U, Leeksma OC, Tomsic R, Feugier P, Salles G, Gabarre J, Kersten MJ, Van Den Neste E, Creemers GJ, Gaillard I, Meijnders P, Tertian G, Reman O, Muller HP, Troncy J, Blanc M, Schroyens W, Voogt PJ, Wijermans P, Rieux C, Ferme C, Henry-Amar M; EORTC-GELA H8 Trial Group. Quality of life after successful treatment of early-stage Hodgkin's lymphoma: 10-year follow-up of the EORTC-GELA H8 randomised controlled trial. Lancet Oncol. 2009 Dec;10(12):1160-70. doi: 10.1016/S1470-2045(09)70258-X. Epub 2009 Oct 12. PMID 19828373
- [Result] Mounier N, Heutte N, Flechtner H, et al.: Quality of life in early stage Hodgkin lymphoma (HL) patients from the EORTC-GELA H8 Trial (20931): A post-treatment longitudinal study of 1,015 patients. [Abstract] J Clin Oncol 26 (Suppl 15): A-9535, 2008.
- [Result] Ferme C, Eghbali H, Meerwaldt JH, Rieux C, Bosq J, Berger F, Girinsky T, Brice P, van't Veer MB, Walewski JA, Lederlin P, Tirelli U, Carde P, Van den Neste E, Gyan E, Monconduit M, Divine M, Raemaekers JM, Salles G, Noordijk EM, Creemers GJ, Gabarre J, Hagenbeek A, Reman O, Blanc M, Thomas J, Vie B, Kluin-Nelemans JC, Viseu F, Baars JW, Poortmans P, Lugtenburg PJ, Carrie C, Jaubert J, Henry-Amar M; EORTC-GELA H8 Trial. Chemotherapy plus involved-field radiation in early-stage Hodgkin's disease. N Engl J Med. 2007 Nov 8;357(19):1916-27. doi: 10.1056/NEJMoa064601. PMID 17989384